CLINICAL TRIAL: NCT00269074
Title: Safety and Efficacy of IDEA-070 for the Treatment of Pain and Inflammation Induced by Photodynamic Therapy of Actinic Keratosis
Brief Title: Effect of IDEA-070 on Pain and Inflammation Induced by PDT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IDEA AG (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CL-070-II-02; EudrCT number: 2005-002875-34
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2009-03-20 (Estimated); Status verified 2009-03

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

INTERVENTIONS:
Drug: IDEA-070

SUMMARY:
Primary objectives: effect of IDEA-070 compared to placebo on pain and inflammation induced by PDT. The primary objective is to detect a statistically significant difference of pain and inflammation induced by PDT in test areas treated with IDEA-070 compared to placebo-treated areas.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis ot actinic keratosis to be treated with PDT affecting equal sized areas of both sides of the head affecting at least 10% of the area of photoexposure

Exclusion Criteria:

Morpheaform basal cell carcinoma, Major hypertrophy of lesions, Porphyria, Topical treatment with 5-FU, cryotherapy, PDT, diclophenac sodium, and other less common treatments on the treatment area or systemic treatment within 3 month prior to screening, Concomitant use of other analgesics including topical NSAIDs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2006-01; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Julia Reifenberger, PD Dr. med., Principal Investigator — Dermatological department of university Duesseldorf
Locations (1):
- Dermatological department of university hospital, Düsseldorf, North Rhine-Westphalia, Germany